CLINICAL TRIAL: NCT06574854
Title: Effects of Descending Stair Walking on Cardiometabolic Adaptations Among Obese, Untrained Women
Brief Title: Effects of Descending Stair Walking
Acronym: DSW
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Universiti Sains Malaysia (Other)
Collaborators: Ministry of Health, Malaysia (Other Government)
Responsible Party: Principal Investigator, Nazirah Gulam Mohamed, Principal Investigator, Universiti Sains Malaysia
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: USM/JEPeM/PP/23070582
Record Dates: First submitted 2024-08-14; First posted 2024-08-28 (Actual); Last update posted 2026-02-05 (Actual); Status verified 2026-02

CONDITIONS: Obesity
Keywords: body composition; cardiometabolic; stair walking; obesity
MeSH Terms: conditions — Obesity

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- DSW (Experimental): Descending Stair Walking
  Interventions: Other: DSW
- ASW (Active Comparator): Ascending Stair Walking
  Interventions: Other: ASW

INTERVENTIONS:
Other: DSW — Descending Stair Walking
  Other Names: Eccentric Training
  Arms: DSW
Other: ASW — Ascending Stair Walking
  Other Names: Concentric Training
  Arms: ASW

SUMMARY:
The global rise in the prevalence of physical inactivity is major public health concern. Lifestyle-related activities, such as stairs walking, has important public health implications and may represent an alternative approach for those who have difficulty adhering to conventional exercise programs. This two-armed, parallel-group, randomized controlled trial (RCT) aims to assess and compare the effects between the descending stair walking (DSW) and ascending stair walking (ASW) on cardiometabolic health markers, cardiopulmonary capacity, body composition and muscular strength.

This RCT will recruit 16 obese inactive and sedentary females will be randomized using permuted block randomization into two arms: intervention arm, DSW and active comparator arm: ASW in a 1:1 allocation ratio. The participants in the DSW and ASW arms will undergo twice a week stair walking intervention session for 8 weeks. The exercise volume will be gradually increased over 8 weeks by increasing the number of repetitions by two every week for both arms. Borg's scale of perceived exertion (RPE) and visual analogue scale (VAS) will be used to assess subjective intensity of stair walking and pain intensity immediately after each repetition. Assessments will be carried out through two time points, pre-intervention assessment (T0) and immediately after completion of the intervention at 8 weeks (T1). During each assessment, the primary outcome to be assessed includes the cardiometabolic health markers and cardiopulmonary capacity, while the secondary outcomes to be assessed are the body composition and muscular strength. Whereas during the intervention, continuous heart rate and gas consumption will be monitored at week 1 (W1), week 4 (W4) and week 8 (W8) to monitor the intensity of the exercise.

DETAILED DESCRIPTION:
1.2 Research Objectives

1.2.1 General Objective (i) The study compares the impact of the 8-week descending stair walking (DSW) and ascending stair walking (ASW) on cardiometabolic health in obese, untrained women.

1.2.2 Specific Objective

To compare the effect of DSW & ASW on:

(i) cardiometabolic health (fasting plasma glucose, lipid profile, renal profile, cardiorespiratory fitness, resting blood pressure, resting energy expenditure, resting heart rate) (ii) body composition (fat mass, lean body mass, waist circumference, hip circumference, thigh circumference) (iii) muscular fitness & functional capacity (back and leg strength & 6-min walking test)

1.3 Research Design This randomized controlled trial (RCT) is a single-centre, two-armed, parallel-group.

1.4 Research Location This RCT is expected to run for 1 year in the Wellness Hub Timur Laut, Klinik Kesihatan Jalan Angsana Pulau Pinang. Wellness Hub Timur Laut is located in the primary healthcare facility of the Ministry of Health and receives approximately 1,000 clients annually for health screening.

1.5 Sampling Method The sampling method used in this study for recruitment of participants is by purposive sampling. Overweight & obese clients of Wellness Hub Jalan Angsana, Klinik Kesihatan Jalan Angsana Pulau Pinang

1.6 Sample Size Calculation The sample size is estimated based on an effect size of 1.91, an α-level of 0.05, and a power (1-β) of 0.08. A priori sample size analysis (G∗Power 3.1; Düsseldorf, Germany) indicated that 6 participants/ group were necessary. Considering a possible dropout rate of 50%, a sample size of 12 participants/ group is anticipated making it a total of 24 participants.

1.7 Data Collection Procedure Permission to conduct the study in Wellness Hub Timur Laut (WHTL), Pulau Pinang, will be sought. Clients will be recruited from WHLA after agreeing to participate in the study.

1.7.1 Data Collection Technique The researcher will interview and assess participants face-to-face at baseline and 8th weeks and the end of the intervention. Participants will be randomly assigned to the stair-walking intervention. At baseline, a background information questionnaire will be used to obtain respondents' sociodemographic characteristics, occupation, health problems and health-related fitness as part of wellness hub health screening. Body composition, metabolic risk factors and selected physical fitness will be assessed before and after the 8th week of intervention.

1.7.2 Daily Energy Balance Monitoring A logbook will be provided for all participants to record daily calorie intake and physical activity. Two weekdays and one-weekend food logs will be retrieved from the logbook, and the total weekly calorie intake and macronutrients will be calculated using Nutritionist Pro software.

1.7.3 Stair Walking Intervention All participants must complete progressive exercise training using stairs in WHLA over 8 weeks, twice a week. The participants in the DSW arm will ride an elevator from level 1 to level 6, eliminating the concentric impact of walking upstairs. Whereas for the ASW arm, participants will ride an elevator from level 6 to level 1 to eliminate the eccentric impact of walking downstairs. The number of stairs from the first to the sixth floor was 120 (five floors, 24 stairs per floor), and the height of each stair was 18 cm. The walking tempo is approximately 1s per step, thus to descend or ascend 120 stairs, it takes about 2 min 30 sec including steps at the landing. The exercise volume will be gradually increased over 8 weeks by increasing the number of repetitions by two repetitions weekly for both arms (first week, 2 repetitions/ session; 8th week, 16 repetitions/ session; 1 repetition,120 stairs).

This protocol assumes that symptoms of muscle damage, such as delayed-onset muscle soreness (DOMS) and prolonged decreases in muscle function, would be minimal after any sessions. It took approximately 5 min to perform one repetition, including the time used for waiting for and riding on an elevator, and the time taken to perform 16 repetitions was approximately 80 min. Lower limb stretching exercises will be included in the workout's general warming-up and cooling-down phases. Over the 16 sessions, each participant will walk up or down 720 floors, thus 17,424 stairs.

ELIGIBILITY:
Inclusion Criteria:

* Women
* age 18-50-year-old
* BMI 25.0 - 39.9 kg/m2,
* body fat percentage > 30%
* no lower limb orthopaedic injuries
* sedentary lifestyle (regular exercise <1 h per week).

Exclusion Criteria:

* smokers
* taking supplements or medication known to affect REE (such as oral contraceptives),
* severe medical conditions affecting their physical or mental health
* individuals with implanted medical device
* suffer from alcohol or drug abuse and
* trying to conceive/ pregnant or breastfeeding

Ages: 18 Years to 50 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes — Female
Enrollment: 24 (Actual)
Dates: Start 2023-05-01 (Actual); Primary Completion 2025-03-01 (Actual); Study Completion 2025-03-15 (Actual)

PRIMARY OUTCOMES:
Total Cholesterol | 8 weeks
  Changes in Total Cholesterol (mmol/L) from baseline
Low-Density Lipoprotein Cholesterol | 8 weeks
  Changes in Low-Density Lipoprotein Cholesterol (mmol/L) from baseline
High-Density Lipoprotein Cholesterol | 8 weeks
  Changes in High-Density Lipoprotein Cholesterol (mmol/L) from baseline
Trigliceride | 8 weeks
  Changes in Trigliceride (mmol/L) from baseline
Fasting Plasma Glucose | 8 weeks
  Changes in Fasting Plasma Glucose (mmol/L) from baseline
Resting Heart Rate | 8 weeks
  Changes in Resting Heart Rate (beat.min) from baseline
Resting Blood Pressure | 8 weeks
  Changes in Resting Diastolic and Systolic Blood Pressure (mm/Hg) from baseline
Resting Energy Expenditure | 8 weeks
  Changes in Resting Energy Expenditure (kcal/day) from baseline
Alanine Aminotransferase | 8 weeks
  Changes in Alanine Aminotransferase (U/L) from baseline
Alanine Aspartate transaminase | 8 weeks
  Changes in Alanine Aspartate transaminase (U/L) from baseline
Resting energy oxidation | 8 weeks
  Changes in fat and charbohydrate oxidation from baseline

SECONDARY OUTCOMES:
Body Mass | 8 weeks
  Changes in body mass (kg)from baseline
Body Mass Index (BMI) | 8 weeks
  Changes in BMI (kg/m2)from baseline
Percentage body fat | 8 weeks
  Changes in percentage body fat (%) from baseline
Lean Body Mass | 8 weeks
  Changes in lean body mass (kg) from baseline
Waist Circumference | 8 weeks
  Changes in waist circumference (cm) from baseline
Hip Circumference | 8 weeks
  Changes in hip circumference (cm) from baseline
Isometric Muscular Strength | 8 weeks
  Changes in back & leg isometric (kg) from baseline
Cardiorespiratory Capacity-6 Minute Walking Test | 8 weeks
  Changes in distance (m) covered from baseline
Training substrate oxidation | 8 weeks
  Changes in substrate oxidation from week 1 to 8

CONTACTS AND LOCATIONS:
Locations (1):
- Wellness Hub Timur Laut, Pulau Pinang, Ayer Itam, Pulau Pinang, Malaysia

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Chen TC, Hsieh CC, Tseng KW, Ho CC, Nosaka K. Effects of Descending Stair Walking on Health and Fitness of Elderly Obese Women. Med Sci Sports Exerc. 2017 Aug;49(8):1614-1622. doi: 10.1249/MSS.0000000000001267. PMID 28291022
- [Background] Regnersgaard S, Knudsen AK, Lindskov FO, Mratinkovic M, Pressel E, Ingersen A, Dela F. Down stair walking: A simple method to increase muscle mass and performance in 65+ year healthy people. Eur J Sport Sci. 2022 Feb;22(2):279-288. doi: 10.1080/17461391.2020.1856936. Epub 2021 Apr 24. PMID 33241972
- [Background] Chen TC, Huang TH, Tseng WC, Tseng KW, Hsieh CC, Chen MY, Chou TY, Huang YC, Chen HL, Nosaka K. Changes in plasma C1q, apelin and adropin concentrations in older adults after descending and ascending stair walking intervention. Sci Rep. 2021 Sep 3;11(1):17644. doi: 10.1038/s41598-021-96631-x. PMID 34480035
- [Background] Theodorou AA, Panayiotou G, Paschalis V, Nikolaidis MG, Kyparos A, Mademli L, Grivas GV, Vrabas IS. Stair descending exercise increases muscle strength in elderly males with chronic heart failure. BMC Res Notes. 2013 Mar 8;6:87. doi: 10.1186/1756-0500-6-87. PMID 23510560
- [Background] Chow BC, Li S, Zhu X, Jiao J, Quach B, Baker JS, Zhang H. Effects of descending or ascending stair exercise on body composition, insulin sensitivity, and inflammatory markers in young Chinese women with obesity: A randomized controlled trial. J Sports Sci. 2021 Mar;39(5):496-502. doi: 10.1080/02640414.2020.1829362. Epub 2020 Oct 4. PMID 33012244
- [Background] Ainsworth BE, Haskell WL, Herrmann SD, Meckes N, Bassett DR Jr, Tudor-Locke C, Greer JL, Vezina J, Whitt-Glover MC, Leon AS. 2011 Compendium of Physical Activities: a second update of codes and MET values. Med Sci Sports Exerc. 2011 Aug;43(8):1575-81. doi: 10.1249/MSS.0b013e31821ece12. PMID 21681120
- [Background] Bassett DR, Vachon JA, Kirkland AO, Howley ET, Duncan GE, Johnson KR. Energy cost of stair climbing and descending on the college alumnus questionnaire. Med Sci Sports Exerc. 1997 Sep;29(9):1250-4. doi: 10.1097/00005768-199709000-00019. PMID 9309638
- [Background] Paschalis V, Theodorou AA, Panayiotou G, Kyparos A, Patikas D, Grivas GV, Nikolaidis MG, Vrabas IS. Stair descending exercise using a novel automatic escalator: effects on muscle performance and health-related parameters. PLoS One. 2013;8(2):e56218. doi: 10.1371/journal.pone.0056218. Epub 2013 Feb 21. PMID 23437093
- [Background] Chen TC, Tseng WC, Huang GL, Chen HL, Tseng KW, Nosaka K. Superior Effects of Eccentric to Concentric Knee Extensor Resistance Training on Physical Fitness, Insulin Sensitivity and Lipid Profiles of Elderly Men. Front Physiol. 2017 Apr 10;8:209. doi: 10.3389/fphys.2017.00209. eCollection 2017. PMID 28443029
- [Background] Ansari M, Hardcastle S, Myers S, Williams AD. The Health and Functional Benefits of Eccentric versus Concentric Exercise Training: A Systematic Review and Meta-Analysis. J Sports Sci Med. 2023 Jun 1;22(2):288-309. doi: 10.52082/jssm.2023.288. eCollection 2023 Jun. PMID 37293426
- [Background] Touron J, Maisonnave L, Rigaudiere JP, Montaurier C, De Antonio M, Perrault H, Richard R, Capel F. Eccentric and concentric exercises induce different adaptions in adipose tissue biology. J Physiol Biochem. 2023 May;79(2):441-450. doi: 10.1007/s13105-023-00956-2. Epub 2023 Mar 24. PMID 36961725